CLINICAL TRIAL: NCT02166645
Title: Comparison of Prone and Supine Positioning in the Immediate Postextubation Period of Preterm Infants: a Randomized Controlled Trial Protocol
Brief Title: Comparison Between Preterm Infants Who Are Placed on Their Back or Stomach in the Immediate Postextubation Period
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uniao Metropolitana de Educacao e Cultura (Other)
Responsible Party: Principal Investigator, Maria Luiza Caires Comper, Master, Uniao Metropolitana de Educacao e Cultura
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCT
Record Dates: First submitted 2014-06-14; First posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-05

CONDITIONS: Pregnancy Preterm
Keywords: patient positioning; premature infant; mechanical ventilation; airway extubation
MeSH Terms: conditions — Premature Birth | interventions — Prone Position; Supine Position

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prone position (Experimental): Prone position per 48 hours after extubation
  Interventions: Other: Prone position
- Supine position (Active Comparator): Supine position per 48 hours after extubation
  Interventions: Other: Supine position

INTERVENTIONS:
Other: Prone position — Participants of intervention group will be placed in prone position immediately after extubation and positioned over a roll to raise the chest and facilitate diaphragmatic dynamic, with lateralized head and aligned with the trunk, upper and lower limbs flexed and hands near the face, facilitating hand-mouth access.
  Other Names: Ventral decubitus
  Arms: Prone position
Other: Supine position — Participants of control group remain in supine position after extubation and positioned with the head in the midline, with the upper side of the thorax and brought forward and rolls down the legs to promote slight flexion (30-40º) in the hips and knees.
  Other Names: Dorsal decubitus
  Arms: Supine position

SUMMARY:
The purpose of this study is to determine whether patient positioning (prone and supine positioning) contributes to the success of extubation in the immediate postextubation period of preterm infants.

DETAILED DESCRIPTION:
This study is double-blinded randomized controlled trial, whose aim is to compare the proportion of successful extubation of preterm infants immediately after the extubation. Methods: Participants will be recruited from neonatal intensive care unit (NICU) and they will be divided into two groups (supine and prone) and positioned in their respective groups after extubation. A clinical evaluation form and a parameters collection form (respiratory rate, heart rate, saturation of peripheral oxygen, fraction of inspired oxygen and temperature) will be used and filled before extubation and 48 hours after by the professional staff of the NICU. It will be considered a successful extubation all participants who staying extubated for 48 hours after extubation.

ELIGIBILITY:
Inclusion Criteria:

* Newborns less than 37 weeks of gestation age (calculated by doctor using the method of Capurro/Ballard)
* Newborns undergone to invasive mechanical ventilation in the first week of life, for more than 48 hours

Exclusion Criteria:

* Newborns who present malformations and clinical or surgical conditions that preclude the positioning in prone or supine after extubation

Max Age: 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Successful extubation | 48 hours after extubation

SECONDARY OUTCOMES:
Improvement of parameters | 48 hours after extubation
  Improvement of parameters (respiratory rate, heart rate, saturation of peripheral oxygen, fraction of inspired oxygen and temperature)

OTHER OUTCOMES:
Decrease complications of mechanical ventilation | 48 hours after extubation

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luiza Caíres Comper, Master, Principal Investigator — Uniao Metropolitana de Educacao e Cultura
Locations (1):
- Manoel Novaes Hospital, Itabuna, Estado de Bahia, Brazil

REFERENCES:
- [Background] Antunes LC, Rugolo LM, Crocci AJ. [Effect of preterm infant position on weaning from mechanical ventilation]. J Pediatr (Rio J). 2003 May-Jun;79(3):239-44. Portuguese. PMID 14506534
- [Background] Bhat RY, Hannam S, Pressler R, Rafferty GF, Peacock JL, Greenough A. Effect of prone and supine position on sleep, apneas, and arousal in preterm infants. Pediatrics. 2006 Jul;118(1):101-7. doi: 10.1542/peds.2005-1873. PMID 16818554
- [Background] Jarus T, Bart O, Rabinovich G, Sadeh A, Bloch L, Dolfin T, Litmanovitz I. Effects of prone and supine positions on sleep state and stress responses in preterm infants. Infant Behav Dev. 2011 Apr;34(2):257-63. doi: 10.1016/j.infbeh.2010.12.014. Epub 2011 Mar 9. PMID 21392826
- [Background] Oliveira TG, Rego MA, Pereira NC, Vaz LO, Franca DC, Vieira DS, Parreira VF. Prone position and reduced thoracoabdominal asynchrony in preterm newborns. J Pediatr (Rio J). 2009 Sep-Oct;85(5):443-8. doi: 10.2223/JPED.1932. English, Portuguese. PMID 19830358
- [Background] Paiva KCA, Beppu OS. Posição prona. J Bras Pneumol. 2005;31(4):332-340.
- [Background] Richter T, Bellani G, Scott Harris R, Vidal Melo MF, Winkler T, Venegas JG, Musch G. Effect of prone position on regional shunt, aeration, and perfusion in experimental acute lung injury. Am J Respir Crit Care Med. 2005 Aug 15;172(4):480-7. doi: 10.1164/rccm.200501-004OC. Epub 2005 May 18. PMID 15901611
- [Background] Sud S, Friedrich JO, Taccone P, Polli F, Adhikari NK, Latini R, Pesenti A, Guerin C, Mancebo J, Curley MA, Fernandez R, Chan MC, Beuret P, Voggenreiter G, Sud M, Tognoni G, Gattinoni L. Prone ventilation reduces mortality in patients with acute respiratory failure and severe hypoxemia: systematic review and meta-analysis. Intensive Care Med. 2010 Apr;36(4):585-99. doi: 10.1007/s00134-009-1748-1. Epub 2010 Feb 4. PMID 20130832